CLINICAL TRIAL: NCT00138502
Title: The Significance of Funguria In Hospitalized Patients
Brief Title: Funguria in Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 02-050
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2007-10

CONDITIONS: Candidiasis
Keywords: Candidiasis, Funguria
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of the study is to test the hypothesis that a subpopulation of patients with candiduria are at significant risk for disseminated disease and would benefit from treatment, while others are at low risk from complications and therefore require no antifungal therapy.

DETAILED DESCRIPTION:
This protocol will attempt to generate a detailed clinical profile of patients with funguria and identify subgroups of patients with funguria at high risk for candiduria and determine the relative risks for obtaining candiduria. In addition, it will look at identifying subgroups of patients with funguria at high risk for candidemia and identifying subgroups of patients with funguria at high risk for death. Finally, it will attempt to determine if funguria independently predicts fungemia or death. Data will be complemented by surveillance of a comparable population without funguria.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with fungi isolated from the urine of any colony count.
2. Patients seen at either Harbor-UCLA Medical Center or Cedars Sinai Medical Center.

Exclusion Criteria:

1. Persons with a previously positive urine fungal culture during the current hospital admission.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 926
Dates: Start 2001-09-17; Primary Completion 2008-12-08 (Actual); Study Completion 2008-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA Center For Vaccine Research, Torrance, California